CLINICAL TRIAL: NCT01979211
Title: Phase II Trial of Post-operative or Definitive Concurrent Radiation and Cetuximab for Locally Advanced Cutaneous Squamous Cell Carcinoma of the Head and Neck
Brief Title: Post-operative Radiation With Cetuximab for Locally Advanced Cutaneous Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Vinita Takiar, Assistant Professor, Department of Radiation Oncology, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCHN-12-001
Record Dates: First submitted 2013-10-24; First posted 2013-11-08 (Estimated); Results first posted 2022-05-10 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cetuximab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetuximab and Radiation (Experimental): Cetuximab 400 mg/m2 IV over 120 minutes loading dose > 4 days prior to initiation of radiation; Cetuximab 250 mg/m2 IV over 60 minutes weekly weeks 2-7 concurrent with Radiation therapy 60-66 Gy in 2 Gy daily fractions
  Interventions: Drug: Cetuximab; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Cetuximab — 400 mg/m2 IV over 120 minutes week 1; 250 mg/m2 IV over 60 minutes weekly weeks 2-7
  Other Names: Erbitux
Radiation: Radiation Therapy — Radiation Therapy 60-66 Gy in 2 Gy fractions starting week 2 of Cetuximab

SUMMARY:
The standard treatment of surgery followed by radiation therapy can stop tumors from growing in the head and neck region in most patients. However, the cancer can recur or can spread to other parts of the body. Cetuximab is a drug that may delay or prevent tumor growth by blocking certain cellular chemical pathways that lead to tumor development. It was approved by the United States Food and Drug Administration (FDA) in 2006 for the treatment of head and neck cancer.

The purpose of this study is to determine how easily cetuximab can be added to treatment with radiation therapy in patients with cutaneous cancer of the head and neck. This study will also look at how well cetuximab added to radiation therapy works over time and how well this treatment is tolerated.

DETAILED DESCRIPTION:
This is a Phase II trial to characterize the feasibility of treating patients with locally advanced cutaneous squamous cell carcinomas of the head and neck with post-operative radiotherapy and cetuximab. Cetuximab has previously been given safely in conjunction with head and neck radiotherapy for mucosal squamous cell carcinoma in multiple phase III trials, and so Phase I data is not necessary here.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically) proven diagnosis of cutaneous squamous cell carcinoma of the head and neck
* Clinical stage >/= T3 or >/= N1, M0 including no distant metastases
* Gross total resection of the primary tumor with curative intent must be completed within 7 weeks of registration
* Performance status of 0-1 within 2 weeks prior to registration
* Age >/= 18
* Adequate labs within 2 weeks prior to registration

Exclusion Criteria:

* Prior invasive malignancy unless disease free for a minimum of 3 years; noninvasive cancers (For example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible) are permitted even if diagnosed and treated < 3 years ago. Patients with a history of T1-2, N0, M0 resected differentiated thyroid carcinoma are considered eligible.
* Prior systemic chemotherapy or anti-epidermal growth factor therapy for the study cancer or for a different prior cancer
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-10; Primary Completion 2022-01-19 (Actual); Study Completion 2022-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vinita Takiar, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cetuximab and Radiation
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cetuximab and Radiation
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local Regional Control
Description: The primary endpoint of this study was 2-year locoregional control (LRC), defined as no evidence of recurrent cancer in the tumor bed and/or neck as assessed via clinical exam and imaging. Locoregional control was estimated by the Kaplan-Meier method. The Kaplan-Meier method is a statistical method used to assess survival times while factoring for censored observations (those who had LRC) and the time for them to be censored.
Time Frame: 2 years
Population: 24 data points were included in the Kaplan-Meier method and yielded an predicted percentage of individuals with LRC at a 2 year mark. Analysis yielded a predicted 91% of subjects had LRC. Extrapolating this percentage to the overall number of participants analyzed, 21.84 subjects had LRC.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Cetuximab and Radiation
Number analyzed (Participants) | 24
percentage of subjects | 91.1 [80 to 100]

2. Secondary Outcome: Percentage of Participants With Disease-free Survival
Description: The primary endpoint of this study was 2-year disease-free survival (DFS), which was the absence of locoregional recurrence or metastatic disease (biopsied when possible). DFS was estimated by the Kaplan-Meier method. The Kaplan-Meier method is a statistical method used to assess survival times while factoring for censored observations (those who were alive disease-free) and the time for them to be censored.
Time Frame: 2 years
Population: 24 data points were included in the Kaplan-Meier method and yielded an predicted percentage of individuals with DFS at a 2 year mark. Analysis predicted 70.8% of subjects were alive with no disease. Extrapolating this percentage to the overall number of participants analyzed, 16.99 subjects were alive with no disease.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab and Radiation
Number analyzed (Participants) | 24
percentage of participants | 70.8 [54.8 to 91.6]

3. Secondary Outcome: Percentage of Participants With Overall Survival
Description: The primary endpoint of this study was 5-year overall survival (OS), defined as the absence of death from any cause during those respective time periods. OS was estimated by the Kaplan-Meier method. The Kaplan-Meier method is a statistical method used to assess survival times while factoring for censored observations (those who were alive) and the time for them to be censored.
Time Frame: 5 years
Population: 24 data points were included in the Kaplan-Meier method and yielded an predicted percentage of individuals with OS at a 5 year mark. Analysis predicted 56.1% of subjects were alive. Extrapolating this percentage to the overall number of participants analyzed, 13.34 subjects were alive at the 5 year mark.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab and Radiation
Number analyzed (Participants) | 24
percentage of participants | 56.1 [38.7 to 81.3]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was followed up to 5 years after the start of treatment. Serious Adverse Events and Other (Not Including Serious) Adverse Events were followed up to 24 months after the start of treatment.
Description: The definition does not differ from clinicialtrials.gov's definitions.
Arm/Group | Cetuximab and Radiation
All-Cause Mortality (participants affected / at risk) | 9/24
Serious Adverse Events (participants affected / at risk) | 3/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab and Radiation (N=24)
Dizziness (Nervous system disorders) | 1 (1)
Lip pain (Gastrointestinal disorders) | 1 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab and Radiation (N=24)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (9)
Alkaline phosphatase increased (Investigations) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (3)
Anemia (Blood and lymphatic system disorders) | 1 (4)
Anorexia (Metabolism and nutrition disorders) | 5 (28)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (11)
Chills (General disorders) | 1 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (3)
Confusion (Psychiatric disorders) | 1 (6)
Constipation (Gastrointestinal disorders) | 3 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (12)
Creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 6 (34)
Diarrhea (Gastrointestinal disorders) | 2 (4)
Dry mouth (Gastrointestinal disorders) | 5 (21)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (21)
Dysgeusia (Nervous system disorders) | 7 (40)
Dysphagia (Gastrointestinal disorders) | 1 (4)
Ear pain (Ear and labyrinth disorders) | 1 (3)
Eye disorders - Other, specify (Eye disorders) | 2 (21)
Eye infection (Eye disorders) | 1 (3)
Eye pain (Eye disorders) | 1 (12)
Facial nerve disorder (Nervous system disorders) | 1 (11)
Facial pain (General disorders) | 3 (5)
Fatigue (General disorders) | 14 (91)
Fever (General disorders) | 1 (2)
Headache (Nervous system disorders) | 3 (23)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (27)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (7)
Infections and infestations - Other, specify (Investigations) | 2 (14)
Infusion related reaction (General disorders) | 1 (7)
Insomnia (Psychiatric disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 13 (81)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (13)
Nausea (Gastrointestinal disorders) | 6 (28)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (4)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (12)
Oral pain (Gastrointestinal disorders) | 3 (18)
Pain (General disorders) | 2 (13)
Pharyngitis (Infections and infestations) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (18)
Rash acneiform (Skin and subcutaneous tissue disorders) | 22 (177)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (7)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (21)
Thromboembolic event (Vascular disorders) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (13)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3)
Upper respiratory infection (Infections and infestations) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 1 (6)
Weight loss (Investigations) | 1 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-03): https://cdn.clinicaltrials.gov/large-docs/11/NCT01979211/Prot_SAP_000.pdf